CLINICAL TRIAL: NCT03084835
Title: Smoking Cessation in Lung Cancer Screening: Integrated Digital/Clinical Approach
Brief Title: Low Dose Computed Tomography for Lung Cancer Screening
Acronym: LDCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Study Accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Truth Initiative (Other)
Responsible Party: Principal Investigator, Ivana Croghan, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-004891; 1R01CA207048-01 (NIH)
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Smoking
Keywords: tobacco; smoking; low dose computed tomography; lung screening; text messaging
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UC (Active Comparator): Usual Care
  Interventions: Behavioral: Usual Care
- WEB+TXT (Active Comparator): Digital Intervention
  Interventions: Behavioral: WEB+TXT
- WEB+TXT+TTS (Active Comparator): Digital plus Counseling Intervention
  Interventions: Behavioral: WEB+TXT+TTS

INTERVENTIONS:
Behavioral: Usual Care — Brief cessation counseling
  Arms: UC
Behavioral: WEB+TXT — Access to Become an Ex website plus text messaging
  Arms: WEB+TXT
Behavioral: WEB+TXT+TTS — Access to Become an Ex website plus text messaging plus consult with a trained tobacco treatment specialist
  Arms: WEB+TXT+TTS

SUMMARY:
This study will evaluate the impact of a proactive, EHR-supported enrollment strategy that links LDCT-eligible smokers with an evidence-based intervention comprised of a web-based program and integrated text messaging. The goal is to provide actionable findings about how to most effectively and cost efficiently promote abstinence in LDCT clinics.

DETAILED DESCRIPTION:
Using a 3-arm randomized trial design with repeated measures at 1, 3, 6, and 12 months, the study will randomize N=1650 smokers who present for LDCT lung cancer screening to an passive referral usual care control condition, proactive referral to a digital cessation intervention that combines web and text messaging, or proactive referral to a digital cessation intervention combined with Tobacco Treatment Specialist counseling. The Study will examine overall effectiveness of the interventions in promoting abstinence, the impact of proactive referral to treatment, and the total cost and cost effectiveness of the interventions. The Study will also examine the representativeness of the enrolled sample and explore barriers and facilitators to intervention adoption with LDCT clinic leaders. The trial is structured as a practical clinical trial to answer key questions of direct relevance to LDCT decision-makers.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for LDCT screening
2. Current smoking (every day/some days)
3. At least weekly use of the Internet
4. Current ownership of cell phone with a text messaging plan
5. Willing to receive study text messages.
6. Ability to complete all aspects of the study
7. Ability to provide signed informed consent

Exclusion Criteria:

1. Current (in the past 30 days) use of tobacco cessation medication or participation in tobacco cessation treatment.
2. Those with a condition deemed by the investigators to be exclusionary to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | 12 months
  biochemically confirmed 12 month smoking abstinence of WEB+TXT;
smoking abstinence | 12 months
  biochemically confirmed 12 month smoking abstinence of WEB+TXT+TTS ;
smoking abstinence | 12 months
  biochemically confirmed 12 month smoking abstinence of UC;

CONTACTS AND LOCATIONS:
Overall Officials: James T Hays, MD, Principal Investigator — Mayo Clinic; David E Midthun, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham AL, Burke MV, Jacobs MA, Cha S, Croghan IT, Schroeder DR, Moriarty JP, Borah BJ, Rasmussen DF, Brookover MJ, Suesse DB, Midthun DE, Hays JT. An integrated digital/clinical approach to smoking cessation in lung cancer screening: study protocol for a randomized controlled trial. Trials. 2017 Nov 28;18(1):568. doi: 10.1186/s13063-017-2312-x. PMID 29179734
- [Background] Burke, MV; Graham, AL; Midthun, DE; Hays, JT; Efficacia delle nuove tecnologie digitali di rete per la smoking cessation nello screening del tumore polmonare (Effectiveness of new digital technologies for smoking cessation in lung cancer screening). Tabaccologia 2019; 2:21-25